CLINICAL TRIAL: NCT06701747
Title: Development and Validation of a Nomogram Predicting the Risk of Perioperative High-dose Transfusion in Non-cardiac Surgery
Brief Title: A Nomogram Predicting the Risk of High-dose Transfusion in Non-cardiac Surgery
Status: Completed | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Ren Liao, Associate professor, West China Hospital
Other Study IDs: WCH20231634
Record Dates: First submitted 2024-11-15; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Massive Transfusion; Nomogram Model
Keywords: Massive transfusion; Red blood cells; Nomogram; Non-cardiac surgery; Patient blood management

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- High-dose group: Receive RBCs transfusion over 1600mL
- No-high-dose group: Receive RBCs transfusion under 1600mL

SUMMARY:
This retrospective study was designed to develop a preoperative nomogram, validated both internally and externally, to supply an individual and precise tool for predicting the probability that patients will require perioperative transfusion therapy.

DETAILED DESCRIPTION:
Perioperative red blood cells (RBCs) transfusion is a necessary guarantee for surgical surgery and one of the indispensable means in modern medical treatment. In recent years, with the continuous improvement of medical standards, various major and complex surgeries have been carried out. The total number of patients receiving surgical treatment increased year by year, and the demand for surgical blood has also increased rapidly. Although unpaid blood donation has been vigorously advocated in recent years, the supply of blood products are still difficult to meet the growing demand for clinical blood. RBCs transfusion is often associated with unavoidable complications such as anaphylaxis and transfusion-related acute lung injury, which may lead to delayed recovery, increased hospital stay and medical costs, and result in serious adverse effects and even death.

Hemorrhage is a common complication of surgery. The effect of blood transfusion treatment and the patient's recovery process will be affected by the amount of blood transfused during the perioperative period. Similarly, blood products that are prepared in advance for surgery often remains unused perioperatively, leading to the waste of valuable blood resources and an increase in hospital expenses. Hemorrhage is one of the leading causes of death in various clinical situations, such as severe trauma, heart surgery, and traffic accidents.Timely and effective high-dose transfusion is directly related to life and death. However, high-dose transfusion may also lead to dilution coagulopathy, increased risk of bleeding, and imbalance in the internal environment.

In brief, there is an urgent requirement for a systematic, evidence-driven tool to comprehensively weigh the risks and benefits of high-dose RBCs transfusion in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing non-cardiac surgery during hospitalization.
* Patients receiving allogeneic RBCs transfusion within 24 hours during and after surgery.

Exclusion Criteria:

* Age under 15 years.
* Patients with incomplete clinical data.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This retrospective study included 【】patients who received RBCs transfusion during non-cardiac surgery at West China Hospital between January 2018 and June 2024.
Sampling Method: Non-Probability Sample
Enrollment: 11197 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
RBCs transfusion volume | Up to 24 hours after transfusion
  The total volume of RBCs transfused within 24 from the start of transfusion.

CONTACTS AND LOCATIONS:
Overall Officials: Ren Liao, M.D., Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No